CLINICAL TRIAL: NCT01879163
Title: A Phase I Randomised Trial to Evaluate the Safety and Immunogenicity of MVA85A-IMX313 Compared to MVA85A in Bacille Calmette-Guérin (BCG) Vaccinated Adults
Brief Title: Phase I Trial Evaluating Safety and Immunogenicity of MVA85A-IMX313 Compared to MVA85A in BCG Vaccinated Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Imaxio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TB028
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Tuberculosis (TB)
Keywords: Vaccine; Immunogenicity
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): The first six volunteers will receive an intradermal injection of 1x10^7 pfu MVA85A-IMX313 (non-randomised).
  Interventions: Biological: MVA85A-IMX313
- Group B (Active Comparator): 12 subjects receiving intradermal injection of 5x10^7 pfu MVA85A-IMX313 (following completion of group A, subjects will be randomised to either group B or group C).
  Interventions: Biological: MVA85A-IMX313
- Group C (Active Comparator): 12 subjects receiving intradermal injection of 5x10^7 pfu MVA85A (following completion of group A, subjects will be randomised to either group B or group C).
  Interventions: Biological: MVA85A

INTERVENTIONS:
Biological: MVA85A-IMX313 — Intradermal injection of MVA85A-IMX313 (MVA85A-IMX313 combines the candidate TB vaccine MVA85A with the carrier protein IMX313)
  Arms: Group A; Group B
Biological: MVA85A — Intradermal injection of MVA85A (recombinant Modified Vaccinia virus Ankara expressing the M. tb antigen 85A)
  Other Names: AERAS-485
  Arms: Group C

SUMMARY:
This is a Phase I trial to evaluate the safety and immunogenicity of MVA85A-IMX313 vaccination compared to MVA85A vaccination, in BCG vaccinated adults.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the trial:

* Healthy adult aged 18-55 years
* Resident in or near Oxford (for CCVTM) or Birmingham (for WTCRF) and able to travel to Oxford for vaccination for the duration of the trial period
* No relevant findings in medical history or on physical examination
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected trial vaccination date (by visible BCG scar on examination or written documentation)
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register subject details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

Subjects must meet none of the following criteria to enter the trial:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with candidate vaccine MVA85A or candidate vaccine FP85A or any other recombinant MVA vaccine
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), autoimmune disease, cancer (except BCC or CIS), cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine, including eggs
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the subject in the trial
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during trial period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the trial vaccine for 30 days prior to dosing with the trial vaccine, or planned use during the trial period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluation through actively and passively collected data on adverse events | Up to 24 weeks
  To evaluate the safety in healthy BCG-vaccinated subjects of MVA85A-IMX313 vaccination compared to MVA85A vaccination, by actively and passively collecting data on adverse events.

SECONDARY OUTCOMES:
Evaluation of immune response of MVA85A-IMX313 vaccination compared with MVA85A vaccination in healthy, BCG vaccinated adults. | Up to 24 weeks
  To evaluate the immune response in healthy BCG-vaccinated subjects of MVA85A-IMX313 vaccination, compared with MVA85A vaccination, by comparing laboratory markers of cell mediated immunity in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire
  - Wellcome Trust Clinical Research Facility, Birmingham

REFERENCES:
- [Derived] Minhinnick A, Satti I, Harris S, Wilkie M, Sheehan S, Stockdale L, Manjaly Thomas ZR, Lopez-Ramon R, Poulton I, Lawrie A, Vermaak S, Le Vert A, Del Campo J, Hill F, Moss P, McShane H. A first-in-human phase 1 trial to evaluate the safety and immunogenicity of the candidate tuberculosis vaccine MVA85A-IMX313, administered to BCG-vaccinated adults. Vaccine. 2016 Mar 8;34(11):1412-21. doi: 10.1016/j.vaccine.2016.01.062. Epub 2016 Feb 5. PMID 26854906
- See also: Jenner Institute, University of Oxford, Website — http://www.jenner.ac.uk/clinicaltrials